CLINICAL TRIAL: NCT02598297
Title: A Randomized, Double Blind, Placebo-controlled, Multicenter, Phase III Study Investigating the Efficacy and Safety of Ruxolitinib in Early Myelofibrosis Patients With High Molecular Risk Mutations
Brief Title: Phase III Study Investigating the Efficacy and Safety of Ruxolitinib in Early Myelofibrosis Patients With High Molecular Risk Mutations.
Acronym: ReTHINK
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unresolvable inability to recruit the patients.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CINC424A2353; 2014-004928-21 (EudraCT Number)
Record Dates: First submitted 2015-10-27; First posted 2015-11-05 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Myelofibrosis With High Molecular Risk Mutations
Keywords: Early Myelofibrosis; high molecular risk mutations.; Ruxolitinib; INC424; High molecular risk mutations; HMR
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib (Active Comparator): Two tablets of ruxolitinib 5 mg were administered orally twice per day.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib Placebo (Placebo Comparator): Two tablets of 5mg placebo were administered orally twice per day.
  Interventions: Drug: Ruxolitinib Placebo

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg tablet for oral use
  Other Names: INC424
  Arms: Ruxolitinib
Drug: Ruxolitinib Placebo — 5 mg placebo tablet for oral use
  Arms: Ruxolitinib Placebo

SUMMARY:
Myelofibrosis patients with high molecular risk mutations have an intrinsically aggressive disease with increased risk of leukemic transformation and reduced overall survival. As there are no therapies currently established in the subset of high molecular risk patients with early myelofibrosis, the study aimed to evaluate ruxolitinib in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MF with bone marrow fibrosis of at least Grade 1; irrespective of JAK2 mutational status
* Patients with at least one mutation in one of the five HMR genes (ASXL1, EZH2, SRSF2 and IDH1/2)
* Patients with non-palpable spleen or spleen palpable ≤ 5 cm from the left costal margin to the point of greatest splenic protrusion
* Patients with MF-7 score of ≤ 15, with each individual symptom score of ≤ 3

Exclusion Criteria:

* Patients with prior treatment with ruxolitinib or other JAK inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (106):
- Australia (4):
  - Novartis Investigative Site, Concord NSW, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Brazil (2):
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Novartis Investigative Site, Toronto, Ontario, Canada
- Denmark (2):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Herlev
- France (9):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Chambéry
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (15):
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Halle S
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nordhorn
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Ulm
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
- Israel (5):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Zrifin
- Italy (12):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Varese, VA
- Japan (10):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Chūō, Yamanashi
  - Novartis Investigative Site, Osaka
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Loerenskog
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Wroclaw
- Portugal (2):
  - Novartis Investigative Site, Faro
  - Novartis Investigative Site, Porto
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Madrid
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Huddinge
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Uddevalla
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- Taiwan (4):
  - Novartis Investigative Site, Putzu City, Chiayi Hsien
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Samsun
  - Novartis Investigative Site, Talas / Kayseri
- United Kingdom (5):
  - Novartis Investigative Site, Edgbaston, Birmingham
  - Novartis Investigative Site, Westbruy on Trym, Bristol
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 320 male or female adults (age 18 or over) with a confirmed diagnosis of MF were planned to be enrolled. The target population was not met due to early study termination. A total of 49 subjects were enrolled in the study, 25 in the ruxolitinib arm and 24 in the placebo arm.
Groups:
- Ruxolitinib (INC424): Two tablets of ruxolitinib 5 mg were administered orally twice per day
Period: Overall Study
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Started | 25 (One subject in the ruxolitinib arm was not treated with the study drug) | 24
Not Treted Wit Study Drug | 1 | 0
Subjects Followed for Survival | 1 | 0
Completed | 0 | 0
Not Completed | 25 | 24
Not completed — Study terminated by Sponsor | 21 | 23
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Subject/guardian decision | 1 | 0
Not completed — Followed for survival | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment.
  Years | 59.0 (14.23) | 67.4 (7.72) | 63.1 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment.
  Participants
    Female | 12 | 7 | 19
    Male | 13 | 17 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment.
  Participants
    Caucasian | 19 | 23 | 42
    Asian | 4 | 1 | 5
    Other | 1 | 0 | 1
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS-1)
Description: Progression free survival (PFS-1) from date of randomization until the occurrence of any of the criteria for disease progression:
  * Progressive splenomegaly
  * Circulating peripheral blast counts > 10%
  * Leukemic transformation
  * Hb < 10g/dl with absolute decrease of at least 3 g/dl from baseline
  * White blood cell (WBC) counts > 25 x 103/ μL
  * MF-7 score ≥ 30
  * Death from any cause
Time Frame: From randomization till disease progression (estimated to be assessed up 48 months)
Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment. This endpoint was not analyzed as study was terminated and it was specified in the statistical analysis plan (SAP) that the primary endpoint of PFS and any other time to event endpoint would not be derived.
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Primary Progression (TTP)
Description: TTP is defined as time from randomization until disease progression as defined for PFS-1 excluding death as an event.
Time Frame: From randomization till progression (estimated to be assessed up to 48 months)
Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment. This endpoint was not analyzed as study was terminated and it was specified in the statistical analysis plan (SAP) that any time to event endpoint would not be derived.
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage Change in Spleen Volume From Baseline
Description: Change in spleen volume (by MRI/CT) from baseline
Time Frame: From baseline and assessed on 12 week intervals until end of treatment (EOT)
Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 25 | 24
Percentage change from baseline
  Week 12: number analyzed (Participants) | 19 | 19
  Week 12 | -10.8 (24.45) | 9.1 (12.34)
  Week 24: number analyzed (Participants) | 13 | 8
  Week 24 | -17.8 (18.83) | 17.6 (17.78)
  Week 36: number analyzed (Participants) | 7 | 2
  Week 36 | -18.4 (31.62) | 32.5 (18.81)
  Week 48: number analyzed (Participants) | 2 | 0
  Week 48 | -23.5 (10.57) |
  End of Treatment (EOT): number analyzed (Participants) | 10 | 9
  End of Treatment (EOT) | -11.6 (8.08) | 18.1 (18.58)

4. Secondary Outcome: Percentage Change in Symptoms From Baseline Using MF-7
Description: Percentage change from Baseline in MF-7 total symptom score and 7 individual symptoms at each visit was summarized with descriptive statistics. For this scale, symptoms range from 0 to 10 for the severity experienced within the past 24 hours, with 0 being for absence of symptoms and 10 for worst imaginable symptoms.
Time Frame: From Baseline and assessed every 4 weeks until end of treatment
Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment.
Measure: Mean (Standard Deviation); unit: Percentage change in scores
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 25 | 24
Percentage change in scores
  Total Score derived (TSD): Baseline (BL) | 6.6 (5.17) | 5.9 (5.56)
  TSD change from baseline @ W12: number analyzed (Participants) | 19 | 20
  TSD change from baseline @ W12 | -0.3 (4.45) | 0.5 (6.08)
  TSD change from baseline @ W24: number analyzed (Participants) | 13 | 9
  TSD change from baseline @ W24 | 0.5 (3.71) | -0.8 (6.44)
  TSD change from baseline @ W48: number analyzed (Participants) | 3 | 0
  TSD change from baseline @ W48 | -0.3 (3.06) |
  TSD change from BL @ EOT: number analyzed (Participants) | 15 | 16
  TSD change from BL @ EOT | 1.1 (4.40) | 3.3 (9.53)
  Tiredness: Baseline (BL) | 1.8 (1.45) | 1.5 (1.53)
  Tiredness: change from baseline @ W12: number analyzed (Participants) | 19 | 20
  Tiredness: change from baseline @ W12 | 0.1 (1.47) | 0.4 (1.27)
  Tiredness: change from baseline @ W24: number analyzed (Participants) | 13 | 9
  Tiredness: change from baseline @ W24 | -0.1 (0.76) | 1.1 (2.52)
  Tiredness: change from baseline @ W48: number analyzed (Participants) | 3 | 0
  Tiredness: change from baseline @ W48 | -0.3 (0.58) |
  Tiredness change from BL @ EOT: number analyzed (Participants) | 15 | 16
  Tiredness change from BL @ EOT | 0.8 (1.32) | 1.1 (2.28)
  Filling up quickly when you eat (FUQWYE):BL | 1.0 (1.41) | 0.8 (1.27)
  FUQWYE: change from BL @W12: number analyzed (Participants) | 19 | 20
  FUQWYE: change from BL @W12 | 0.1 (1.49) | -0.1 (2.09)
  FUQWYE: change from BL @W24: number analyzed (Participants) | 13 | 9
  FUQWYE: change from BL @W24 | -0.2 (0.99) | 0.1 (1.17)
  FUQWYE: change from BL @W48: number analyzed (Participants) | 3 | 0
  FUQWYE: change from BL @W48 | 0.7 (1.15) |
  FUQWYE: change from BL @ EOT: number analyzed (Participants) | 15 | 16
  FUQWYE: change from BL @ EOT | 0.2 (1.08) | 0.3 (2.29)
  Abdominal discomfort (AD): BL | 0.7 (1.43) | 0.6 (1.10)
  Abdominal discomfort change from BL @W12: number analyzed (Participants) | 19 | 20
  Abdominal discomfort change from BL @W12 | -0.1 (1.66) | -0.1 (0.85)
  Abdominal discomfort change from BL @W24: number analyzed (Participants) | 13 | 9
  Abdominal discomfort change from BL @W24 | 0.0 (1.15) | -0.3 (0.71)
  Abdominal discomfort change from BL @W48: number analyzed (Participants) | 3 | 0
  Abdominal discomfort change from BL @W48 | 0.0 (0.00) |
  AD: change from BL @ EOT: number analyzed (Participants) | 15 | 16
  AD: change from BL @ EOT | 0.1 (0.92) | 0.3 (1.40)
  Night sweat (NS): Baseline (BL) | 0.7 (1.07) | 1.1 (1.45)
  Night sweat change from BL @W12: number analyzed (Participants) | 19 | 20
  Night sweat change from BL @W12 | -0.1 (0.71) | -0.3 (1.29)
  Night sweat change from BL @W24: number analyzed (Participants) | 13 | 9
  Night sweat change from BL @W24 | 0.5 (1.45) | -0.7 (1.41)
  Night sweat change from BL @W48: number analyzed (Participants) | 3 | 0
  Night sweat change from BL @W48 | -0.3 (0.58) |
  Night Sweat: change from BL @ EOT: number analyzed (Participants) | 15 | 16
  Night Sweat: change from BL @ EOT | 0.0 (0.85) | 0.3 (2.12)
  Itching (Pruritus):BL | 0.9 (1.42) | 0.6 (0.93)
  Itching (Pruritus): change from BL @W12: number analyzed (Participants) | 19 | 20
  Itching (Pruritus): change from BL @W12 | -0.3 (0.67) | 0.1 (1.45)
  Itching (Pruritus): change from BL @W24: number analyzed (Participants) | 13 | 9
  Itching (Pruritus): change from BL @W24 | 0.4 (0.77) | -0.3 (1.22)
  Itching (Pruritus): change from BL @W48: number analyzed (Participants) | 3 | 0
  Itching (Pruritus): change from BL @W48 | -1.0 (1.73) |
  Itching: change from BL @ EOT: number analyzed (Participants) | 15 | 16
  Itching: change from BL @ EOT | 0.1 (1.03) | 0.4 (1.75)
  Bone Pain: BL | 0.9 (1.35) | 0.9 (1.33)
  Bone Pain: change from BL @W12: number analyzed (Participants) | 19 | 20
  Bone Pain: change from BL @W12 | -0.4 (1.01) | 0.3 (1.56)
  Bone Pain: change from BL @W24: number analyzed (Participants) | 13 | 9
  Bone Pain: change from BL @W24 | -0.2 (1.17) | -0.8 (1.79)
  Bone Pain: change from BL @W48: number analyzed (Participants) | 3 | 0
  Bone Pain: change from BL @W48 | 0.7 (1.15) |
  Bone Pain: change from BL @ EOT: number analyzed (Participants) | 15 | 16
  Bone Pain: change from BL @ EOT | 0.1 (0.96) | 0.6 (1.50)
  Pain under ribs on left side (PUROLS): BL | 0.7 (1.18) | 0.4 (0.82)
  PUROLS: change from BL @W12: number analyzed (Participants) | 19 | 20
  PUROLS: change from BL @W12 | 0.4 (1.01) | 0.1 (0.76)
  PUROLS: change from BL @W24: number analyzed (Participants) | 13 | 9
  PUROLS: change from BL @W24 | 0.0 (0.41) | 0.1 (1.17)
  PUROLS: change from BL @W48: number analyzed (Participants) | 3 | 0
  PUROLS: change from BL @W48 | 0.0 (0.00) |
  PUROLS: change from BL @ EOT: number analyzed (Participants) | 15 | 16
  PUROLS: change from BL @ EOT | -0.2 (0.68) | 0.3 (1.00)

5. Secondary Outcome: Number of Participants With Specific Subscale Scores (From Baseline) Using EQ-5D
Description: EQ-ED5 profiles were summarized at baseline and at each scheduled assessment for each of the 5 dimensions separately (Mobility, self-care, usual activities, pain discomfort, anxiety/depression) Only participants with baseline score and at least one non-missing post-baseline score during the treatment period were included. Percentages were based on all these evaluable participants.
  The 5 scores for mobility, self-care, usual activities, pain/discomfort and anxiety/depression are all self-explanatory (eg "I have no problems walking" to "I am unable to walk"), except for the following overall health check, where 100 is the best of health, and 0 is the worst health.
Time Frame: From Baseline and assessed every 4 weeks until end of treatment
Population: The Full Analysis Set (FAS) included all subjects who were randomized to a study treatment. Only the categories with non-zero counts are presented with these results. Only subjects with baseline score and at least one non-missing post-baseline score during the treatment period 1 were included. % is based on all these evaluable subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 25 | 24
Participants
  Mobility- Baseline: No problem | 17 | 18
  Mobility- Baseline: Slight problems | 4 | 5
  Mobility- Baseline: Moderate problems | 1 | 1
  Mobility- Baseline: Extreme problems | 1 | 0
  Mobility - Week 4:No prob. | 17 | 14
  Mobility - Week 4: Slight problems | 4 | 7
  Mobility - Week 4: Moderate problems | 1 | 2
  Mobility - Week 8: No problem | 17 | 15
  Mobility - Week 8: Slight problems | 3 | 6
  Mobility - Week 8: Moderate problems | 0 | 1
  Mobility - Week 12: No problem | 15 | 12
  Mobility - Week 12: Slight problems | 4 | 6
  Mobility - Week 12: Moderate problems | 0 | 2
  Mobility - Week 16: No problem | 12 | 10
  Mobility - Week 16: Slight problems | 2 | 7
  Mobility - Week 16: Moderate problems | 1 | 0
  Mobility - Week 20: No problem | 12 | 5
  Mobility - Week 20: Slight problems | 2 | 6
  Mobility - Week 24: No problem | 12 | 5
  Mobility - Week 24: Slight problems | 1 | 3
  Mobility - Week 24: Moderate problems | 0 | 1
  Mobility - Week 32: No problem | 8 | 1
  Mobility - Week 32: Slight problems | 0 | 1
  Mobility - Week 32: Moderate problems | 1 | 0
  Mobility - Week 40: No problem | 5 | 0
  Mobility - Week 40: Slight problems | 1 | 0
  Mobility - Week 48: No problem | 2 | 0
  Mobility - Week 48: Slight problems | 1 | 0
  Mobility - EOT: No problem | 11 | 12
  Mobility - EOT: Slight problems | 4 | 3
  Mobility - EOT: Moderate problems | 0 | 1
  Mobility- 30 day safety FU: No problem | 2 | 3
  Mobility- 30 day safety FU: Slight problems | 1 | 0
  Self-care - Baseline: No problem | 23 | 22
  Self-care - Baseline: Slight problems | 0 | 2
  Self-care - Week 4: No problem | 21 | 20
  Self-care - Week 4: Slight problems | 0 | 3
  Self-care - Week 4: Moderate problems | 1 | 0
  Self-care - Week 8: No problem | 19 | 21
  Self-care - Week 8: Slight problems | 1 | 1
  Self-care - Week 12: No problem | 17 | 19
  Self-care - Week 12: Slight problems | 1 | 1
  Self-care - Week 12: Moderate problems | 1 | 0
  Self-care - Week 16: No problem | 15 | 16
  Self-care - Week 16: Slight problems | 0 | 1
  Self-care - Week 20: No problem | 14 | 11
  Self-care - Week 24: No problem | 12 | 9
  Self-care - Week 24: Slight problems | 1 | 0
  Self-care - Week 32: No problem | 8 | 2
  Self-care - Week 32: Slight problems | 1 | 0
  Self-care - Week 40: No problem | 5 | 0
  Self-care - Week 40: Slight problems | 1 | 0
  Self-care - Week 48: No problem | 3 | 0
  Self-care - EOT: No problem | 14 | 15
  Self-care - EOT: Slight problems | 1 | 1
  Self-care - 30 day Safety FU: No problem | 3 | 3
  Usual activities -Baseline: No problem | 18 | 21
  Usual activities -Baseline: Slight problems | 4 | 3
  Usual activities - Baseline: Moderate problems | 1 | 0
  Usual activities - Week 4: No problem | 20 | 18
  Usual activities - Week 4: Slight problems | 1 | 4
  Usual activities - Week 4: Moderate problems | 1 | 0
  Usual activities - Week 4: Severe problems | 0 | 1
  Usual activities - Week 8: No problem | 20 | 18
  Usual activities - Week 8: Slight problems | 0 | 3
  Usual activities - Week 8: Moderate problems | 0 | 1
  Usual activities - Week 12: No problem | 16 | 16
  Usual activities - Week 12: Slight problems | 3 | 3
  Usual activities - Week 12: Moderate problems | 0 | 1
  Usual activities - Week 16: No problem | 13 | 14
  Usual activities - Week 16: Slight problems | 2 | 3
  Usual activities - Week 20: No problem | 13 | 9
  Usual activities - Week 20: Slight problems | 1 | 2
  Usual activities - Week 24: No problem | 12 | 9
  Usual activities - Week 24: Slight problems | 1 | 0
  Usual activities - Week 32: No problem | 8 | 2
  Usual activities - Week 32: Slight problems | 1 | 0
  Usual activities - Week 40: No problem | 5 | 0
  Usual activities - Week 40: Slight problems | 1 | 0
  Usual activities - Week 48: No problem | 3 | 0
  Usual activities - EOT: No problem | 12 | 13
  Usual activities -EOT: Slight problems | 3 | 3
  Usual activities - 30 day Safety FU: No problem | 2 | 3
  Usual activities - 30 say Safety FU: Slight probs | 1 | 0
  Pain/Discomfort - Baseline: No problem | 13 | 11
  Pain/Discomfort - Baseline: Slight problems | 8 | 12
  Pain/Discomfort - Baseline: Moderate problems | 2 | 1
  Pain/Discomfort - Week 4: No problem | 11 | 15
  Pain/Discomfort - Week 4: Slight problems | 10 | 6
  Pain/Discomfort - Week 4: Moderate problems | 1 | 2
  Pain/Discomfort - Week 8: No problem | 14 | 13
  Pain/Discomfort - Week 8: Slight problems | 5 | 7
  Pain/Discomfort - Week 8: Moderate problems | 1 | 2
  Pain/Discomfort - Week 12: No problem | 12 | 10
  Pain/Discomfort - Week 12: Slight problems | 7 | 6
  Pain/Discomfort - Week 12: Moderate problems | 0 | 4
  Pain/Discomfort - Week 16: No problem | 9 | 11
  Pain/Discomfort - WK16: Slight problems | 6 | 3
  Pain/Discomfort - WK16: Moderate problems | 0 | 3
  Pain/Discomfort - WK20: No problem | 8 | 8
  Pain/Discomfort - WK20: Slight problems | 6 | 3
  Pain/Discomfort - WK24: No problem | 9 | 7
  Pain/Discomfort - WK24: Slight problems | 4 | 2
  Pain/Discomfort - WK32: No problem | 7 | 2
  Pain/Discomfort - WK32: Slight problems | 2 | 0
  Pain/Discomfort - WK40: No problem | 4 | 0
  Pain/Discomfort - WK40: Slight problems | 2 | 0
  Pain/Discomfort - WK48: No problem | 3 | 0
  Pain/Discomfort - EOT: No problem | 8 | 10
  Pain/Discomfort - EOT: Slight problems | 7 | 3
  Pain/Discomfort - EOT: Moderate problems | 0 | 3
  Pain/Discomfort - 30 day Safety FU: No problem | 1 | 2
  Pain/Discomfort - 30 day safety FU: Slight probs | 2 | 0
  Pain/Discomfort - 30 day Safety FU: Moderate probs | 0 | 1
  Anxiety/Depression - Baseline: No problem | 14 | 18
  Anxiety/Depression - Baseline: Slight problems | 6 | 3
  Anxiety/Depression - Baseline: Moderate problems | 3 | 3
  Anxiety/Depression - WK4: No problem | 13 | 15
  Anxiety/Depression - WK4: Slight problems | 7 | 6
  Anxiety/Depression - WK4: Moderate problems | 2 | 2
  Anxiety/Depression - WK8: No problem | 11 | 16
  Anxiety/Depression - WK8: Slight problems | 8 | 2
  Anxiety/Depression - WK8: Moderate problems | 1 | 4
  Anxiety/Depression - WK12: No problem | 8 | 13
  Anxiety/Depression - WK12: Slight problems | 10 | 3
  Anxiety/Depression -WK12: Moderate problems | 1 | 4
  Anxiety/Depression - WK16: No problem | 10 | 10
  Anxiety/Depression - WK16: Slight problems | 5 | 5
  Anxiety/Depression - WK16: Moderate problems | 0 | 2
  Anxiety/Depression -WK20: No problem | 10 | 8
  Anxiety/Depression - WK20: Slight problems | 4 | 3
  Anxiety/Depression - WK24: No problem | 11 | 7
  Anxiety/Depression - WK24: Slight problems | 2 | 2
  Anxiety/Depression - WK32: No problem | 7 | 2
  Anxiety/Depression - WK32: Slight problems | 2 | 0
  Anxiety/Depression - WK40: No problem | 5 | 0
  Anxiety/Depression - WK40: Slight problems | 1 | 0
  Anxiety/Depression - WK48: No problem | 3 | 0
  Anxiety/Depression - EOT: No problem | 11 | 12
  Anxiety/Depression - EOT: Slight probs | 4 | 3
  Anxiety/Depression - EOT: Moderate probs | 0 | 1
  Anxiety/Depression - 30 day Safety FU: No probs | 2 | 2
  Anxiety/Depression-30 day Safety FU: Slight probs | 1 | 0
  Anxiety/Depression-30 day Safety FU: Severe probs | 0 | 1

6. Secondary Outcome: Overall Survival
Description: To evaluate the effect of ruxolitinib on overall survival
Time Frame: Time from randomization to date of death due to any cause (estimated to be assessed up to 48 months).
Population: as for outcome 2
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Plasma Ruxolitinib Concentrations
Description: Characterize pharmacokinetics (PK)by utilizing a population PK approach.
Time Frame: Week 12, Wk 48
Population: The Pharmacokinetics (PK) Analysis Set (PAS) consisted of all patients set who have received at least one dose of ruxolitinib and provided evaluable PK data. The PK analysis was never done as the study terminated early.
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Progression Free Survival (PFS-2)
Description: PFS-2 assessed by 25% increase over new baseline of PFS-1 in any of the following: ● Progressive splenomegaly ● 25 % increase in MF-7 score with absolute score ≥ 30
Time Frame: From date of randomization until second disease progression or death, whichever comes first (estimated to be assessed up to 72 months)
Population: as for outcome 2
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Quality-adjusted Life Years From Baseline
Description: EQ-5D-5L (EuroQol-5D-5L, is a standardized instrument for measuring health outcomes, is consists of a descriptive system and a visual analogue scale - scores can be summarized into a single index score that provides a simple measure of health for clinical and economic appraisal ) The EQ-5D-5L health states will be converted into index values (utilities) from which the QALY (Quality - adjusted life years) will be calculated. QALY will be summarized descriptively by treatment arm.
Time Frame: Change from Baseline compared with scheduled study visits at the following intervals every 4 weeks up to week 24, every 8 weeks up to Week 48, every 12 weeks past Wk 48 until End of treatment and 30 day follow up visit
Population: as for outcome 2
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Time to First Progressive Splenomegaly (TTPS)
Description: Time to first progressive splenomegaly as determined by spleen volume (by Magnetic Resonance Imaging (MRI)/Computed Tomography (CT).
Time Frame: From randomization until earliest time to progressive splenomegaly (estimated to be assessed up to 48 months)
Population: as for outcome 2
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to First Symptomatic Progression (TTSP)
Description: Time to first symptomatic progression as determined by Myelofibrosis 7 Item Symptom Scale (MF-7)
Time Frame: From randomization until symptomatic progression (MF-7)(estimated to be assessed up to 48 months)
Population: as for outcome 2
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately up to approx. 55.1 weeks.
Description: One subject in the ruxolitinib arm was not treated with the study drug due to subject or guardian's decision post randomization. This subject is included in the FAS but not in the Safety set.
Arm/Group | Ruxolitinib (INC424) | Ruxolitinib Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/24
Other Adverse Events (participants affected / at risk) | 17/24 | 11/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (INC424) (N=24) | Ruxolitinib Placebo (N=24)
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (INC424) (N=24) | Ruxolitinib Placebo (N=24)
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Fatigue (General disorders) | 3 | 4
Pyrexia (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2015-09-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT02598297/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT02598297/SAP_001.pdf